CLINICAL TRIAL: NCT02446912
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Phase 3 Study Evaluating the Efficacy and Safety of Two Doses of Anifrolumab in Adult Subjects With Active Systemic Lupus Erythematosus
Brief Title: Efficacy and Safety of Two Doses of Anifrolumab Compared to Placebo in Adult Subjects With Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3461C00005
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Active Systemic Lupus Erythematosus
Keywords: Active Systemic Lupus Erythematosus
MeSH Terms: interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Anifrolumab - higher dose (Experimental): Anifrolumab
  Interventions: Biological: Anifrolumab
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Anifrolumab - lower dose (Experimental): Anifrolumab
  Interventions: Biological: Anifrolumab

INTERVENTIONS:
Biological: Anifrolumab — Anifrolumab IV administration every 4 weeks from Week 0 to Week 48 for a total of 13 doses
  Arms: Anifrolumab - higher dose; Anifrolumab - lower dose
Drug: Placebo — Placebo IV administration every 4 weeks from Week 0 to Week 48
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an intravenous treatment regimen of two doses of anifrolumab versus placebo in adult subjects with moderately to severely active, autoantibody-positive systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is a Phase 3, multicentre, multinational, randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of an intravenous treatment regimen of two doses of anifrolumab versus placebo in subjects with moderately to severely active, autoantibody-positive systemic lupus erythematosus (SLE) while receiving standard of care (SOC) treatment. The study will be performed in adult subjects aged 18 to 70 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 through 70 years at the time of screening
2. Diagnosis of paediatric or adult SLE with a diagnosis of SLE according to the ACR 1982 revised criteria ≥24 weeks prior to signing the Informed Consent form (ICF)
3. Currently receiving at least 1 of the following:

   1. Where prednisone is the single standard of care medication (ie, the subject is not concurrently receiving any medication listed in inclusion criterion 3(c)), a dose of oral prednisone ≥7.5 mg/day but ≤40 mg/day (or prednisone equivalent) for a minimum of 8 weeks prior to Day 1. In addition, the dose of oral prednisone or prednisone equivalent the subject is taking must be stable for a minimum of 2 weeks prior to randomisation.
   2. Where prednisone is not the single standard of care medication (ie, the subject is concurrently receiving at least one medication listed in inclusion criterion 3(c)), a dose of oral prednisone (≤40 mg/day) (or prednisone equivalent) for a minimum of 2 weeks prior to signing of the ICF. In addition, the dose of oral prednisone or prednisone equivalent the subject is taking must be stable for a minimum of 2 weeks prior to randomisation.
   3. Any of the following medications administered for a minimum of 12 weeks prior to signing the informed consent, and at a stable dose for a minimum of 8 weeks prior to signing the informed consent through Day 1:

   (i) Azathioprine ≤200 mg/day (ii) Antimalarial (eg, chloroquine, hydroxychloroquine, quinacrine) (iii) Mycophenolate mofetil ≤2 g/day or mycophenolic acid ≤1.44 g/day (iv) Oral, subcutaneous (SC), or intramuscular methotrexate ≤25 mg/week (v) Mizoribine ≤150 mg/day
4. Fulfils at least 4 of the 11 ACR modified 1982 classification criteria for SLE, at least 1 of which must be:

   1. Positive antinuclear antibody (ANA) test at screening by immunofluorescent assay (IFA) at the central laboratory with titre ≥1:80; OR
   2. Anti-dsDNA antibodies at screening elevated to above normal (including indeterminante), as per the central laboratory; OR
   3. Anti-Smith (anti-Sm) antibody at screening elevated to above normal as per the central laboratory.
5. At Screening, Disease Activity Adjudication Group confirmation of:

   SLEDAI-2K Criteria: SLEDAI-2K score ≥6 points and "Clinical" SLEDAI-2K score ≥4 points. The "Clinical" SLEDAI-2K is the SLEDAI-2K assessment score without the inclusion of points attributable to any urine or laboratory results including immunologic measures.
6. Must not have active or latent TB on either chest radiograph or by quantiferon gold test
7. Day 1 "Clinical" SLEDAI-2K score ≥4 points
8. OCS dose stable for at least 2 weeks prior to randomisation
9. Stable SLE SOC treatment at the time of randomisation
10. Women of child-bearing potential must have a negative serum β-hCG test and negative urine pregnancy test at randomisation (Day 1) prior to administration of investigational product

Exclusion Criteria:

1. Receipt of any investigational product (small molecule or biologic agent) within 4 weeks or 5 half-lives prior to signing of the ICF, whichever is greater
2. Receipt of any of the following:

   (a) Intra-articular, intramuscular or IV glucocorticosteroids within 6 weeks prior to Day 1
3. History of, or current diagnosis of, a clinically significant non SLE-related vasculitis syndrome.
4. Active severe or unstable neuropsychiatric SLE
5. Active severe SLE-driven renal disease
6. Diagnosis (within 1 year of signing the ICF) of mixed connective tissue disease or any history of overlap syndromes of SLE or SSc.
7. History of, or current, inflammatory joint or skin disease other than SLE
8. History of any non-SLE disease that has required treatment with oral or parenteral corticosteroids for more than 2 weeks within the last 24 weeks prior to signing the ICF
9. Known history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the subject to infection, or a positive result for human immunodeficiency virus (HIV) infection confirmed by central laboratory at screening. Subjects refusing HIV testing during the screening period will not be eligible for study participation
10. Confirmed positive test for hepatitis B or hepatitis C
11. Any severe herpes infection at any time prior to Week 0 (Day 1)
12. Opportunistic infection requiring hospitalisation or intravenous antimicrobial treatment within 3 years prior to randomization
13. History of cancer, apart from:

    1. Squamous or basal cell carcinoma of the skin that has been successfully treated
    2. Cervical cancer in situ that has been successfully treated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Hutman, MD, Study Director — Medical Science Director
Locations (122):
- United States (45):
  - Research Site, Birmingham, Alabama
  - Research Site, El Cajon, California
  - Research Site, La Jolla, California
  - Research Site, Los Alamitos, California
  - Research Site, Thousand Oaks, California
  - Research Site, Aurora, Colorado
  - Research Site, Aventura, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Plantation, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Idaho Falls, Idaho
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Hagerstown, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Nashua, New Hampshire
  - Research Site, Freehold, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Jackson, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Glendale, Wisconsin
- Argentina (2):
  - Research Site, Córdoba
  - Research Site, San Miguel de Tucumán
- Australia (3):
  - Research Site, Fitzroy
  - Research Site, Kogarah
  - Research Site, St Leonards
- Brazil (4):
  - Research Site, Belo Horizonte
  - Research Site, Juiz de Fora
  - Research Site, Porto Alegre
  - Research Site, Salvador
- Chile (3):
  - Research Site, Osorno
  - Research Site, Santiago
  - Research Site, Viña del Mar
- Colombia (5):
  - Research Site, Armenia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Medellín
- Germany (6):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dessau-RoBlau
  - Research Site, Frankfurt am Main
  - Research Site, Göttingen
  - Research Site, Kirchheim
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
  - Research Site, Zalaegerszeg
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
- Italy (2):
  - Research Site, Milan
  - Research Site, Padua
- New Zealand (2):
  - Research Site, Hamilton
  - Research Site, Wellington
- Peru (2):
  - Research Site, Arequipa
  - Research Site, Lima
- Poland (12):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Nadarzyn
  - Research Site, Poznan
  - Research Site, Sosnowiec
  - Research Site, Starachowice
  - Research Site, Szczecin
  - Research Site, Ustroń
  - Research Site, Warsaw
- Romania (5):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Galati
  - Research Site, Tg Mures
- South Korea (5):
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Suwon
- Taiwan (3):
  - Research Site, Kaohsiung Hsien
  - Research Site, Taichung
  - Research Site, Taipei
- Ukraine (7):
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (7):
  - Research Site, Brighton
  - Research Site, Doncaster
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Romford
  - Research Site, Staffordshire

REFERENCES:
- [Derived] Furie RA, Morand EF, Bruce IN, Manzi S, Kalunian KC, Vital EM, Lawrence Ford T, Gupta R, Hiepe F, Santiago M, Brohawn PZ, Berglind A, Tummala R; TULIP-1 study investigators. Type I interferon inhibitor anifrolumab in active systemic lupus erythematosus (TULIP-1): a randomised, controlled, phase 3 trial. Lancet Rheumatol. 2019 Dec;1(4):e208-e219. doi: 10.1016/S2665-9913(19)30076-1. Epub 2019 Nov 11. PMID 38229377
- [Derived] Morand EF, Abreu G, Furie RA, Golder V, Tummala R. Lupus low disease activity state attainment in the phase 3 TULIP trials of anifrolumab in active systemic lupus erythematosus. Ann Rheum Dis. 2023 May;82(5):639-645. doi: 10.1136/ard-2022-222748. Epub 2023 Jan 23. PMID 36690388
- [Derived] Bruce IN, van Vollenhoven RF, Morand EF, Furie RA, Manzi S, White WB, Abreu G, Tummala R. Sustained glucocorticoid tapering in the phase 3 trials of anifrolumab: a post hoc analysis of the TULIP-1 and TULIP-2 trials. Rheumatology (Oxford). 2023 Apr 3;62(4):1526-1534. doi: 10.1093/rheumatology/keac491. PMID 36018235
- [Derived] Bruce IN, Furie RA, Morand EF, Manzi S, Tanaka Y, Kalunian KC, Merrill JT, Puzio P, Maho E, Kleoudis C, Albulescu M, Hultquist M, Tummala R. Concordance and discordance in SLE clinical trial outcome measures: analysis of three anifrolumab phase 2/3 trials. Ann Rheum Dis. 2022 Jul;81(7):962-969. doi: 10.1136/annrheumdis-2021-221847. Epub 2022 May 17. PMID 35580976
- [Derived] Vital EM, Merrill JT, Morand EF, Furie RA, Bruce IN, Tanaka Y, Manzi S, Kalunian KC, Kalyani RN, Streicher K, Abreu G, Tummala R. Anifrolumab efficacy and safety by type I interferon gene signature and clinical subgroups in patients with SLE: post hoc analysis of pooled data from two phase III trials. Ann Rheum Dis. 2022 Jul;81(7):951-961. doi: 10.1136/annrheumdis-2021-221425. Epub 2022 Mar 25. PMID 35338035
- [Derived] Loncharich MF, Anderson CW. Interferon Inhibition for Lupus with Anifrolumab: Critical Appraisal of the Evidence Leading to FDA Approval. ACR Open Rheumatol. 2022 Jun;4(6):486-491. doi: 10.1002/acr2.11414. Epub 2022 Feb 14. PMID 35157371
- [Derived] Chia YL, Zhang J, Tummala R, Rouse T, Furie RA, Morand EF. Relationship of anifrolumab pharmacokinetics with efficacy and safety in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2022 May 5;61(5):1900-1910. doi: 10.1093/rheumatology/keab704. PMID 34528084
- [Derived] Furie R, Morand EF, Askanase AD, Vital EM, Merrill JT, Kalyani RN, Abreu G, Pineda L, Tummala R. Anifrolumab reduces flare rates in patients with moderate to severe systemic lupus erythematosus. Lupus. 2021 Jul;30(8):1254-1263. doi: 10.1177/09612033211014267. Epub 2021 May 12. PMID 33977796
- [Derived] Furie R, Morand EF, Bruce IN, Isenberg D, van Vollenhoven R, Abreu G, Pineda L, Tummala R. What Does It Mean to Be a British Isles Lupus Assessment Group-Based Composite Lupus Assessment Responder? Post Hoc Analysis of Two Phase III Trials. Arthritis Rheumatol. 2021 Nov;73(11):2059-2068. doi: 10.1002/art.41778. Epub 2021 Sep 22. PMID 33913260
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: CSP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00005&attachmentIdentifier=dbb257f6-3341-4f6e-87e5-8cef8eb24694&fileName=CSP_D3461C00005_redacted.pdf&versionIdentifier=
- See also: SAP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00005&attachmentIdentifier=fbbb0a3a-88f7-446c-81fe-9e642be982ce&fileName=SAP_D3461C00005_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the trial at 123 sites in 18 countries worldwide.
Groups:
- Anifrolumab 150 mg: Anifrolumab (150 mg) administered via an intravenous infusion (IV) every 4 weeks for up to 48 weeks (13 doses)
- Anifrolumab 300 mg: Anifrolumab (300 mg) administered via an intravenous infusion (IV) every 4 weeks for up to 48 weeks (13 doses)
- Placebo: Matching placebo administered via an intravenous infusion (IV) every 4 weeks for up to 48 weeks (13 doses)
Period: Overall Study
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Started | 93 | 180 | 184
Participants Who Completed Week 52 | 80 | 153 | 157
Completed | 75 | 145 | 149
Not Completed | 18 | 35 | 35
Not completed — Adverse Event | 3 | 13 | 5
Not completed — Condition under investigation worsened | 0 | 1 | 1
Not completed — Study-specific withdrawal criteria | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 4 | 7
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Severe non-compliance to protocol | 1 | 0 | 1
Not completed — Withdrawal by Subject | 10 | 15 | 15
Not completed — Miscellaneous | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo | Total
Number analyzed (Participants) | 93 | 180 | 184 | 457
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (12.05) | 42.0 (11.99) | 41.0 (12.30) | 41.3 (12.11)
Age, Customized [Count of Participants; unit: Participants]
  < 18 | 0 | 0 | 0 | 0
  ≥ 18 to < 65 | 90 | 169 | 178 | 437
  ≥ 65 | 3 | 11 | 6 | 20
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
  Participants
    Female | 86 | 165 | 171 | 422
    Male | 7 | 15 | 13 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
  Participants
    Hispanic or Latino | 20 | 32 | 35 | 87
    Not Hispanic or Latino | 73 | 148 | 149 | 370
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
  Participants
    American Indian or Alaska Native | 0 | 0 | 1 | 1
    Asian | 8 | 11 | 5 | 24
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 14 | 29 | 23 | 66
    White | 64 | 125 | 137 | 326
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 7 | 15 | 18 | 40
Height [Mean (Standard Deviation); unit: cm] — Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
  cm | 164.02 (8.208) | 162.99 (7.829) | 163.10 (8.030) | 163.24 (7.980)
Weight [Mean (Standard Deviation); unit: kg] — Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
  kg | 73.57 (19.469) | 75.36 (20.343) | 74.69 (19.332) | 74.72 (19.731)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
  kg/m2 | 27.31 (6.81) | 28.25 (6.899) | 28.09 (7.145) | 28.00 (6.976)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Systemic Lupus Erythematosus (SLE) Responder Index ≥4 (SRI[4]) at Week 52 (Original Analysis With Restricted Medication Rules)
Description: SRI(4) was defined as meeting all of the following criteria:
  Reduction from baseline of ≥4 points in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) No new organ systems affected, defined by 1 or more British Isles Lupus Assessment Group (BILAG-2004) A or 2 or more BILAG-2004 B items No worsening from baseline in participants lupus disease activity. Worsening was defined as an increase of ≥0.30 points on a 3-point Physician's Global Assessment (PGA) visual analogue scale (VAS) No discontinuation of investigational product and no use of restricted medications beyond the pre-specified analysis threshold.
Time Frame: Week 52
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 35 | 65 | 74
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — The difference in estimates and associated 95% CI are weighted and are calculated using a stratified Cochran-Mantel-Haenszel (CMH) approach, with stratification factors (SLEDAI-2K score at screening [<10 points vs >= 10 points], Week 0 OCS dose [<10 mg/day vs >=10 mg/day prednisone or equivalent] and type I IFN gene signature test result at screening [high vs low]); p = 0.412, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-14.2 to 5.8]
Statistical Analysis 2: Comparison: Anifrolumab 150 mg vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-14.7 to 9.6]

2. Post Hoc Outcome: Number of Participants Who Achieved a Systemic Lupus Erythematosus (SLE) Responder Index ≥4 (SRI[4]) at Week 52 (Post-Hoc Analysis With Revised Restricted Medication Rules)
Description: SRI(4) was defined as meeting all of the following criteria:
  Reduction from baseline of ≥4 points in the SLEDAI-2K No new organ systems affected, defined by 1 or more BILAG-2004 A or 2 or more BILAG-2004 B items No worsening from baseline in lupus disease activity. Worsening defined as an increase of ≥0.30 points on a 3-point PGA VAS No discontinuation of investigational product and no use of restricted medications beyond the revised post-hoc allowed threshold.
  Revised rules were designed to be more clinically appropriate, capture intent of protocol, minimize the risk of restricted medications confounding efficacy, and to allow appropriate quantification and interpretation of the relevant endpoints.
Time Frame: Week 52
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 45 | 84 | 79
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.455, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-6.3 to 14.1]
Statistical Analysis 2: Comparison: Anifrolumab 150 mg vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-6.7 to 17.8]

3. Secondary Outcome: Number of Participants Who Achieved a Systemic Lupus Erythematosus (SLE) Responder Index of ≥4 at Week 52 in the Interferon (IFN) Test-High Sub-Group (Original Analysis With Restricted Medication Rules)
Description: SRI(4) was defined as meeting all of the following criteria:
  Reduction from baseline of ≥4 points in the SLEDAI-2K No new organ systems affected, defined by 1 or more BILAG-2004 A or 2 or more BILAG-2004 B No worsening from baseline in participants lupus disease activity. Worsening was defined as an increase of ≥0.30 points on a 3-point PGA VAS No discontinuation of investigational product and no use of restricted medications beyond the pre-specified analysis threshold.
Time Frame: Week 52
Population: All participants who received investigational product with non-missing baseline measurements, and high IFN test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 76 | 148 | 151
Participants | 30 | 53 | 59
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.549, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-14.4 to 7.6]

4. Post Hoc Outcome: Number of Participants Who Achieved an Systemic Lupus Erythematosus (SLE) Responder Index of ≥4 at Week 52 in the Interferon (IFN) Test-High Sub-Group (Post-Hoc Analysis With Revised Restricted Medication Rules)
Description: SRI(4) was defined as meeting all of the following criteria:
  Reduction from baseline of ≥4 points in the SLEDAI-2K No new organ systems affected, defined by 1 or more BILAG-2004 A or 2 or more BILAG-2004 B items No worsening from baseline in lupus disease activity. Worsening defined as an increase of ≥0.30 points on a 3-point PGA VAS No discontinuation of investigational product and no use of restricted medications beyond the revised post-hoc analysis threshold.
  Revised rules were designed to be more clinically appropriate, capture intent of protocol, minimize the risk of restricted medications confounding efficacy, and to allow appropriate quantification and interpretation of the relevant endpoints.
Time Frame: Week 52
Population: All participants who received investigational product with non-missing baseline measurements, and high IFN test results.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 76 | 148 | 151
Participants | 40 | 71 | 63
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.261, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [-4.8 to 17.7]

5. Secondary Outcome: Number of Participants Who Achieved and Maintained an Oral Corticosteroid (OCS) Dose of ≤7.5 mg/Day in the Sub-group of Participants With Baseline OCS ≥10 mg/Day (Original Analysis With Restricted Medication Rules)
Description: Maintained OCS reduction was defined by meeting all the following criteria:
  Achieve an OCS dose of ≤7.5 mg/day prednisone or equivalent by Week 40 Maintain an OCS dose ≤7.5 mg/day prednisone or equivalent from Week 40 to Week 52 No discontinuation of investigational product and no use of restricted medications beyond the pre-specified analysis threshold.
Time Frame: Week 52
Population: All participants who received investigational product, who had a baseline OCS ≥10 mg/day, and had non-missing baseline measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 48 | 103 | 102
Participants | 17 | 42 | 33
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.180, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 8.9, 95% CI 2-sided [-4.1 to 21.9]

6. Post Hoc Outcome: Number of Participants Who Achieved and Maintained an Oral Corticosteroid (OCS) Dose of ≤7.5 mg/Day in the Sub-group of Participants With Baseline OCS ≥10 mg/Day (Post-Hoc Analysis With Revised Restricted Medication Rules)
Description: Maintained OCS reduction was defined by meeting all of the following criteria:
  Achieve an OCS dose of ≤7.5 mg/day prednisone or equivalent by Week 40 Maintain an OCS dose ≤7.5 mg/day prednisone or equivalent from Week 40 to Week 52 No discontinuation of investigational product and no use of restricted medications beyond the revised post-hoc analysis threshold.
  Revised rules were designed to be more clinically appropriate, capture intent of protocol, minimize the risk of restricted medication confounding efficacy, and to allow appropriate quantification and interpretation of the relevant endpoints.
Time Frame: Week 52
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 48 | 103 | 102
Participants | 24 | 50 | 33
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.013, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 16.7, 95% CI 2-sided [3.5 to 29.8]

7. Secondary Outcome: Number of Participants With a ≥50% Reduction in CLASI Activity Score at Week 12 in the Sub-group of Participants With Baseline CLASI Activity Score ≥10 (Original Analysis With Restricted Medication Rules)
Description: 50% reduction in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score compared to baseline was defined by meeting all of the following criteria:
  Achieve ≥50% reduction of CLASI activity score at Week 12 compared to baseline No discontinuation of investigational product and no use of restricted medications beyond the pre-specified analysis threshold before assessment.
Time Frame: Week 12
Population: All participants who received investigational product, had a baseline CLASI Activity Score ≥10, and had non-missing baseline measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 30 | 58 | 54
Participants | 15 | 24 | 14
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.054, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 17.0, 95% CI 2-sided [-0.3 to 34.3]

8. Post Hoc Outcome: Number of Participants With a ≥50% Reduction in CLASI Activity Score at Week 12 in the Sub-group of Participants With Baseline CLASI Activity Score ≥10 (Post-Hoc Analysis With Revised Restricted Medication Rules)
Description: 50% reduction in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score compared to baseline was defined by meeting all the following criteria:
  Achieve ≥50% reduction of CLASI activity score at Week 12 compared to baseline No discontinuation of investigational product and no use of restricted medications beyond the revised post-hoc analysis threshold before assessment.
  Revised rules were designed to be more clinically appropriate, capture intent of protocol, minimize the risk of restricted medication confounding efficacy, and to allow appropriate quantification and interpretation of the relevant endpoints.
Time Frame: Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 30 | 58 | 54
Participants | 16 | 25 | 14
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.034, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 18.7, 95% CI 2-sided [1.4 to 36.0]

9. Secondary Outcome: Number of Participants Who Achieved a Systemic Lupus Erythematosus (SLE) Responder Index of ≥4 (SRI[4]) at Week 24 (Original Analysis With Restricted Medication Rules)
Description: SRI(4) was defined as meeting all of the following criteria:
  Reduction from baseline of ≥4 points in the SLEDAI-2K No new organ systems affected as defined by 1 or more BILAG-2004 A or 2 or more BILAG-2004 B items No worsening from baseline in participants lupus disease activity. Worsening was defined as an increase of ≥0.30 points on a 3-point PGA VAS No discontinuation of investigational product and no use of restricted medications beyond the pre-specified threshold.
Time Frame: Week 24
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 34 | 74 | 75
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.905, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-9.4 to 10.6]

10. Post Hoc Outcome: Number of Participants Who Achieved a Systemic Lupus Erythematosus (SLE) Responder Index of ≥4 (SRI[4]) at Week 24 (Post-Hoc Analysis With Revised Restricted Medication Rules)
Description: as for outcome 2
Time Frame: Week 24
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 40 | 83 | 79
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.515, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-6.7 to 13.4]

11. Secondary Outcome: Annualized Flare Rate
Description: A flare was defined as either 1 or more new British Isle Lupus Assessment Group (BILAG-2004) A or 2 or more new BILAG-2004 B items compared to the previous visit. The occurrence of a new flare was checked for each available visit versus the previous available visit up to Week 52. If no new flares occurred, the number of flares was set to 0. Otherwise all flares were counted leading to the maximum number of flares of 13. The annualized flare rate was calculated as the number of flares divided by the flare exposure time in days multiplied with 365.25 (1 year). The flare exposure time is the time up to Week 52 (date of BILAG-2004 assessment at Week 52) or up to the date of last available BILAG-2004 assessment.
Time Frame: Baseline to Week 52
Population: Full analysis set - all randomized participants who received investigational product with non-missing baseline measurements.
Measure: Number; unit: Annualized flare rate ratio
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Annualized flare rate ratio | 0.62 | 0.60 | 0.72
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — Analysed using a negative binomial regression model. The response variable in the model is the number of flares over the 52-week treatment period. The model includes covariates of treatment group, and the stratification factors (SLEDAI-2K score at screening [<10 points vs >=10 points], Week 0 OCS dose [<10 mg/day vs >=10 mg/day prednisone or equivalent] and type I IFN gene signature test result at screening [high vs low]). The logarithm of the follow-up time is used as an offset variable; p = 0.258, Negative binomial regression — Nominal p-value; Rate Ratio = 0.83, 95% CI 2-sided [0.60 to 1.14]

12. Secondary Outcome: Number of Participants Who Met the Criteria for British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) Response (Original Analysis With Restricted Medication Rules)
Description: A BICLA responder was achieved if all of the following criteria was met:
  All criteria related to SRI(4) (please see primary endpoint) plus:
  Reduction of all baseline BILAG-2004 A to B/C/D and baseline BILAG-2004 B to C/D, and no BILAG-2004 worsening in other organ systems, as defined by 1 or more BILAG-2004 A or 1 or more new BILAG-2004 B item No discontinuation of investigational product and no use of restricted medications beyond the revised post-hoc analysis threshold before assessment.
Time Frame: Week 52
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 27 | 67 | 49
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [0.6 to 19.7]

13. Post Hoc Outcome: Number of Participants Who Met the Criteria for British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) Response (Post-Hoc Analysis With Revised Restricted Medication Rules)
Description: A BICLA responder was achieved if all of the following criteria was met:
  All criteria related to SRI(4) (please see primary endpoint) plus:
  Reduction of all baseline BILAG-2004 A to B/C/D and baseline BILAG-2004 B to C/D, and no BILAG-2004 worsening in other organ systems, as defined by 1 or more BILAG-2004 A or 1 or more new BILAG-2004 B item No discontinuation of investigational product and no use of restricted medications beyond the revised post-hoc analysis threshold before assessment.
  Revised rules were designed to be more clinically appropriate, capture intent of protocol, minimize the risk of restricted medications confounding efficacy, and to allow appropriate quantification and interpretation of the relevant endpoints.
Time Frame: Week 52
Population: Full analysis set - all randomized participants who received at least one dose of investigation product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 35 | 83 | 54
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 16.4, 95% CI 2-sided [6.7 to 26.2]

14. Secondary Outcome: Number of Participants Reporting One or More Adverse Events (AE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. AEs were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE). The reported value is inclusive of serious and non-serious AEs.
Time Frame: Baseline to End of Trial (Maximum of 60 weeks)
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 80 | 161 | 145

15. Secondary Outcome: Number of Participants Reporting One or More Adverse Events of Special Interest (AESI)
Description: An AESI is an AE of scientific and medical concern specific to understanding biologics and requires close monitoring and rapid communication by the Investigator to the Sponsor/Sponsor's delegate. An AESI may be serious or nonserious. The events of interest are serious infections, including non opportunistic serious infections, opportunistic infections, anaphylaxis, malignancy, herpes zoster, TB (including latent TB), influenza, vasculitis (non-SLE), and MACE (including stroke, MI, or cardiovascular death).
  AEs were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE).
Time Frame: Baseline to End of Trial (Maximum of 60 weeks)
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 11 | 23 | 18

16. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Signs
Description: Vital signs included oral temperature, blood pressure (BP), pulse rate, and respiratory rate.
  Vital signs were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE).
Time Frame: Baseline to End of Trial (Maximum of 60 weeks)
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 14 | 36 | 46

17. Secondary Outcome: Number of Participants With Markedly Abnormal Physical Examinations
Description: Physical examinations included height and weight. Participants were weighed at each study visit and any medically significant changes were reported.
  Physical examination values were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE).
Time Frame: Baseline to End of Trial (Maximum of 60 weeks)
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 3 | 2 | 2

18. Secondary Outcome: Number of Participants With Markedly Abnormal Electrocardiogram (ECG) Scores
Description: ECGs documented the date, time, heart rate, QRS duration, PR interval, RR interval, QT, and corrected QT interval, which were calculated using the Fridericia formula. The investigator judged the overall interpretation as normal or abnormal, and if abnormal it was decided as to whether or not the abnormality was clinically significant or not clinically significant.
Time Frame: Baseline to Week 52
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Mild To Moderate Lupus Flare Evaluated by Modified Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-SLEDAI Flare Index
Description: The modified SELENA flare index was completed by the Investigator or delegated/qualified physician. Assessment of flares were scored in comparison to the participant's previous visit and should only include findings which, in the opinion of the Investigator, are due to systemic lupus erythematosus (SLE) disease activity within that timeframe. Flare was defined as any 1 criterion present in either the Mild/Moderate Flare or Severe Flare categories.
  Number of flares were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE).
Time Frame: Baseline to End of Trial (Maximum of 60 weeks)
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 38 | 58 | 67

20. Secondary Outcome: Number of Participants With Markedly Abnormal Laboratory Tests
Description: Laboratory tests were collected at central clinical laboratories and included hematology, serum chemistry and urinalysis tests. Laboratory values were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE).
Time Frame: Baseline to End of Trial (Maximum of 60 weeks)
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants | 44 | 71 | 87

21. Secondary Outcome: Number of Participants With Suicidal Ideation or Behaviour Assessed Via the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an assessment tool that evaluates suicidal ideation and behavior. Number of participants with suicidal ideation or behavior was defined as the number of participants who answered "yes" at any time during the treatment period (Baseline to Week 52) to one of the 10 categories:
  Category 1: Wish to be dead Category 2: Non-specific active suicidal thoughts Category 3: Active suicidal ideation with any methods (not plan) without intent to act Category 4: Active suicidal ideation with some intent to act, without specific plan Category 5: Active suicidal ideation with specific plan and intent Category 6: Preparatory acts or behavior Category 7: Aborted attempt Category 8: Interrupted attempt Category 9: Actual attempt (non-fatal) Category 10: Completed suicide
Time Frame: Baseline to Week 52
Population: Full analysis set - all randomized participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 93 | 180 | 184
Participants
  Suicidal ideation | 1 | 2 | 2
  Suicidal behaviour | 0 | 0 | 1

22. Secondary Outcome: Change From Baseline in Personal Health Questionnaire Depression Scale-8 (PHQ-8) Score
Description: PHQ-8 is a 8-item self-report scale, all items are rated on a score of 0-3, for a total range of 0-24. PHQ-8 assesses symptoms of depression over the previous 2 weeks. Higher scores indicate more depressive symptoms. A negative change from baseline score indicates improvement in symptoms.
Time Frame: Baseline to Week 52
Population: All participants who received study drug with non-missing baseline and week 52 measurements.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 71 | 130 | 138
Score on a Scale | -2.1 (4.43) | -2.7 (5.58) | -1.7 (5.40)

ADVERSE EVENTS:
Time Frame: Baseline to End of Trial (Maximum of 60 weeks post first dose)
Description: AEs were either spontaneously reported by the participant or reported in response to open questions, revealed by observation, or were changes from baseline/deterioration in tests and vital signs that met SAE criteria or led to IP discontinuation. Full analysis set: All participants who had received at least one dose of investigational product.
Arm/Group | Anifrolumab 150 mg | Anifrolumab 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/93 | 1/180 | 1/184
Serious Adverse Events (participants affected / at risk) | 10/93 | 27/180 | 35/184
Other Adverse Events (participants affected / at risk) | 78/93 | 157/180 | 141/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anifrolumab 150 mg (N=93) | Anifrolumab 300 mg (N=180) | Placebo (N=184)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 2 (2)
Appenicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neuropsychiatric lupus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (6) | 5 (6)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anifrolumab 150 mg (N=93) | Anifrolumab 300 mg (N=180) | Placebo (N=184)
Hypersensitivity (Immune system disorders) | 4 (6) | 11 (12) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 3 (3)
Nasopharyngitis (Infections and infestations) | 15 (18) | 36 (58) | 24 (28)
Upper respiratory tract infection (Infections and infestations) | 17 (25) | 22 (27) | 19 (27)
Urinary tract infection (Infections and infestations) | 8 (10) | 22 (29) | 26 (32)
Bronchitis (Infections and infestations) | 7 (9) | 15 (17) | 9 (11)
Pharyngitis (Infections and infestations) | 6 (8) | 12 (13) | 13 (15)
Herpes zoster (Infections and infestations) | 5 (5) | 10 (10) | 3 (3)
Sinusitis (Infections and infestations) | 5 (6) | 8 (12) | 12 (13)
Pneumonia (Infections and infestations) | 4 (5) | 4 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 5 (5) | 5 (5) | 2 (3)
Oral herpes (Infections and infestations) | 0 (0) | 8 (10) | 5 (8)
Cellulitis (Infections and infestations) | 0 (0) | 6 (6) | 2 (2)
Folliculitis (Infections and infestations) | 4 (5) | 3 (4) | 3 (3)
Conjunctivitis (Infections and infestations) | 2 (2) | 4 (5) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 5 (7) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1) | 4 (9) | 4 (4)
Tooth infection (Infections and infestations) | 0 (0) | 5 (5) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 3 (3) | 4 (4)
Onychomycosis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Furuncle (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (4)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 4 (4)
Hordeolum (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4)
Steroid withdrawal syndrome (Endocrine disorders) | 0 (0) | 5 (5) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 4 (5)
Depression (Psychiatric disorders) | 7 (7) | 6 (8) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (5) | 4 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4) | 8 (9)
Headache (Nervous system disorders) | 6 (8) | 17 (37) | 18 (23)
Migraine (Nervous system disorders) | 4 (4) | 5 (6) | 5 (6)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 7 (8)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 4 (4) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 11 (13) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 6 (9) | 14 (14)
Vomiting (Gastrointestinal disorders) | 4 (7) | 9 (9) | 4 (6)
Nausea (Gastrointestinal disorders) | 3 (5) | 9 (10) | 14 (19)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 5 (5) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 3 (6) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (6) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (5) | 8 (11)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 11 (13) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (10) | 13 (16)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 5 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4)
Renal colic (Renal and urinary disorders) | 0 (0) | 4 (5) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 5 (8) | 4 (5)
Chest pain (General disorders) | 1 (1) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1) | 5 (6)
Fatigue (General disorders) | 0 (0) | 4 (5) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 3 (3)
Peripheral swelling (General disorders) | 2 (2) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 2 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (17) | 16 (37) | 13 (32)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 6 (7) | 4 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02446912/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT02446912/SAP_003.pdf